CLINICAL TRIAL: NCT05223868
Title: A Phase 2b Multicenter, Randomized, Placebo Controlled, Dose-ranging Study to Evaluate the Efficacy and Safety of JNJ-77242113 for the Treatment of Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study of JNJ-77242113 in Participants With Moderate-to-severe Plaque Psoriasis
Acronym: FRONTIER 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109138; 2021-003700-41 (EudraCT Number); 77242113PSO2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: JNJ-77242113 Dose 1 Once Daily (QD) and Placebo (Experimental): Participants will receive JNJ-77242113 Dose 1 QD and placebo from Week 0 through Week 16. Participants will receive placebo to maintain the blinding of dose regimens.
  Interventions: Drug: JNJ-77242113; Drug: Placebo
- Group 2: JNJ-77242113 Dose 2 QD and Placebo (Experimental): Participants will receive JNJ-77242113 Dose 2 QD and placebo from Week 0 through Week 16. Participants will receive placebo to maintain the blinding of dose regimens.
  Interventions: Drug: JNJ-77242113; Drug: Placebo
- Group 3: JNJ-77242113 Dose 3 QD and Placebo (Experimental): Participants will receive JNJ-77242113 Dose 3 QD and placebo from Week 0 through Week 16. Participants will receive placebo to maintain the blinding of dose regimens.
  Interventions: Drug: JNJ-77242113; Drug: Placebo
- Group 4: JNJ-77242113 Dose 1 Twice Daily (BID) and Placebo (Experimental): Participants will receive JNJ-77242113 Dose 1 BID and placebo from Week 0 through Week 16. Participants will receive placebo to maintain the blinding of dose regimens.
  Interventions: Drug: JNJ-77242113; Drug: Placebo
- Group 5: JNJ-77242113 Dose 3 BID and Placebo (Experimental): Participants will receive JNJ-77242113 Dose 3 BID and placebo from Week 0 through Week 16. Participants will receive placebo to maintain the blinding of dose regimens.
  Interventions: Drug: JNJ-77242113; Drug: Placebo
- Group 6: Placebo (Placebo Comparator): Participants will receive placebo BID from Week 0 through Week 16.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-77242113 — JNJ-77242113 tablet will be administered orally.
  Arms: Group 1: JNJ-77242113 Dose 1 Once Daily (QD) and Placebo; Group 2: JNJ-77242113 Dose 2 QD and Placebo; Group 3: JNJ-77242113 Dose 3 QD and Placebo; Group 4: JNJ-77242113 Dose 1 Twice Daily (BID) and Placebo; Group 5: JNJ-77242113 Dose 3 BID and Placebo
Drug: Placebo — Placebo tablet will be administered orally.

SUMMARY:
Th purpose of the study is to evaluate the dose response of JNJ-77242113 in efficacy at Week 16 in participants with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
The populations of people living with moderate to severe psoriasis is approximately 3.5 billion which are mostly managed with topical and conventional therapies. JNJ-77242113, investigational drug, targets the immune responses in the body and skin which impacts diseases, such as psoriasis and psoriatic arthritis (PsA) and this study evaluates JNJ-77242113 as options of advanced therapies in moderate to severe plaque psoriasis. The total duration of this study is up to 24 weeks which includes a screening period of less than or equal to (<=) 4 weeks, a 16-week treatment period, and a 4-week safety follow-up period. Safety will be assessed by adverse events (AEs), clinical safety laboratory assessments, electrocardiograms (ECGs), vital signs and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of plaque psoriasis, with or without psoriatic arthritis (PsA), for at least 6 months prior to the first administration of study intervention
* Participant be a candidate for phototherapy or systemic treatment for plaque psoriasis
* Participant has a total body surface area (BSA) greater than or equal to (>=)10 percent (%) at screening and baseline
* Participant has a total Psoriasis area and severity index (PASI) >=12 at screening and baseline
* Participant has a total Investigator global assessment (IGA) >=3 at screening and baseline

Exclusion Criteria:

* Participant has a nonplaque form of psoriasis (for example, erythrodermic, guttate, or pustular)
* Participant has current drug-induced psoriasis (for example, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Participant have previously received any other therapeutic agent directly targeted to interleukin 23 receptor (IL-23R) (including but not limited to guselkumab, tildrakizumab, or risankizumab)
* Participant has received any therapeutic agent directly targeted to interleukin 17 receptor (IL-17) or interleukin 12/23 receptor (IL-12/23) (including but not limited to secukinumab, ixekizumab, brodalumab, or ustekinumab) or has received anti-tumor necrosis factor [TNF]-alpha biologic therapy (including, but not limited to adalimumab) within 12 weeks or 5 half-lives, whichever is longer, of the first administration of study intervention
* Participant has received agents that deplete B cells (including, but not limited to, rituximab, or alemtuzumab) within 26 weeks of the first administration of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (76):
- United States (21):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Pacific Skin Institute, Sacramento, California
  - Renstar Medical Research, Ocala, Florida
  - Forcare Clinical Research Inc, Tampa, Florida
  - Atlanta Dermatology, Vein & Research Center, Alpharetta, Georgia
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Dawes Fretzin Clinical Research Group LLC, Indianapolis, Indiana
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - DermAssociates, PC, Rockville, Maryland
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Vivida Dermatology, Las Vegas, Nevada
  - Windsor Dermatology, PC, East Windsor, New Jersey
  - Oregon Dermatology and Research Center, Portland, Oregon
  - University of Pittsburgh Department of Dermatology, Pittsburgh, Pennsylvania
  - Modern Research Associates, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Center for Clinical Studies, Webster, Texas
  - Virginia Clinical Research, Norfolk, Virginia
  - Dermatology Associates, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington
- Canada (4):
  - Dermatrials Research, Hamilton, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Innovaderm Research, Montreal, Quebec
- France (3):
  - Centre Hospitalier Le Mans, Le Mans
  - Hopital Charles Nicolle, Rouen
  - HIA Sainte Anne, Toulon
- Germany (14):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charite - Universitaetsmedizin Berlin (CCM), Berlin
  - Rothhaar Studien GmbH, Berlin
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Niesmann & Othlinghaus GbR, Bochum
  - Rosenpark Research GmbH, Darmstadt
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Derma-Study-Center Friedrichshafen GmbH, Friedrichshafen
  - MensingDerma research GmbH, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - Universitatsklinikum Leipzig AOR, Leipzig
  - Dermatologische Gemeinschaftspraxis, Mahlow
  - Hautarztpraxis, Witten
- Japan (10):
  - Yamanashi Prefectural Central Hospital, Kofu
  - Miyata Dermatology Clinic, Matsudo
  - Takagi Dermatological Clinic, Obihiro-shi
  - Kume Clinic, Sakai
  - Sapporo Skin Clinic, Sapporo
  - Shizuoka General Hospital, Shizuoka
  - Shirasaki Dermatology Clinic, Takaoka
  - Kumamoto Kenhoku Hospital, Tamana
  - Toyama Prefectural Central Hospital, Toyama
  - Nomura Dermatology Clinic, Yokohama
- Poland (5):
  - Nzoz Zdrowie Osteo-Medic, Bialystok
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Dermodent Centrum Medyczne Aldona Czajkowska Rafal Czajkowski S C, Osielsko
  - Klinika Ambroziak Estederm Sp. z o.o, Warsaw
  - Wro Medica, Wroclaw
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - KyungHee University Hospital, Seoul
- Spain (5):
  - Hosp. Univ. Germans Trias I Pujol, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Provincial de Pontevedra, Pontevedra
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. de Manises, Valencia
- Taiwan (4):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- United Kingdom (5):
  - Castle Hill Hospital, Cottingham
  - Russell's Hall Hospital, Dudley
  - Guys and St Thomas NHS Foundation Trust, London
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Mid Yorkshire Hospital NHS Trust- Pinderfields Hospital, Wakefield

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Strawn D, Krueger JG, Bissonnette R, Eyerich K, Ferris LK, Paller AS, Pinter A, Richards D, Chen EY, Paget K, Horowitz D, Parast R, Rusbuldt JJ, Sendecki J, Bhagat S, Tomsho LP, Chou CH, Polak ME, Keyes BE, Bozenhardt E, Xiong Y, Zhou W, DeKlotz C, Newbold P, Waterworth DM, Miller M, Ota T, Yang YW, Leung MW, Miller LS, Cuff CA, McRae B, Ruane D, Kannan AK. Icotrokinra induces early and sustained pharmacodynamic responses in phase IIb study of patients with moderate-to-severe psoriasis. JCI Insight. 2025 Dec 22;10(24):e193563. doi: 10.1172/jci.insight.193563. eCollection 2025 Dec 22. PMID 41424381
- [Derived] Bissonnette R, Pinter A, Ferris LK, Gerdes S, Rich P, Vender R, Miller M, Shen YK, Kannan A, Li S, DeKlotz C, Papp K. An Oral Interleukin-23-Receptor Antagonist Peptide for Plaque Psoriasis. N Engl J Med. 2024 Feb 8;390(6):510-521. doi: 10.1056/NEJMoa2308713. PMID 38324484

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants with moderate to severe plaque psoriasis received 2 tablets of placebo matching to JNJ- 77242113 in morning and 1 tablet in the evening to maintain the blind from Week 0 through Week 16. At Week 16 participants had the option to enroll in long-term extension (LTE) study 77242113PSO2002 (NCT05364554). Participants who were not enrolled in LTE study were followed up for safety up to 4 weeks after the last dose of the study drug at Week 16.
- JNJ-77242113 25 mg QD: Participants with moderate to severe plaque psoriasis received JNJ-77242113 25 milligrams (mg) once daily (QD) and matching placebo in morning followed by matching placebo in the evening to maintain the blind from Week 0 through Week 16. At Week 16 participants had the option to enroll in LTE study 77242113PSO2002 (NCT05364554). Participants who were not enrolled in LTE study were followed up for safety up to 4 weeks after the last dose of the study drug at Week 16.
- JNJ-77242113 50 mg QD: Participants with moderate to severe plaque psoriasis received JNJ-77242113 50 mg QD (2*25 mg tablets) in morning followed by matching placebo in the evening to maintain the blind from Week 0 through Week 16. At Week 16 participants had the option to enroll in LTE study 77242113PSO2002 (NCT05364554). Participants who were not enrolled in LTE study were followed up for safety up to 4 weeks after the last dose of the study drug at Week 16.
- JNJ-77242113 25 mg BID: Participants with moderate to severe plaque psoriasis received JNJ-77242113 25 mg twice daily (BID) in morning and evening along with a matching placebo in the morning to maintain the blind from Week 0 through Week 16. At Week 16 participants had the option to enroll in LTE study 77242113PSO2002 (NCT05364554). Participants who were not enrolled in LTE study were followed up for safety up to 4 weeks after the last dose of the study drug at Week 16.
- JNJ-77242113 100 mg QD: Participants with moderate to severe plaque psoriasis received JNJ-77242113 100 mg QD and matching placebo in morning followed by matching placebo in the evening to maintain the blind from Week 0 through Week 16. At Week 16 participants had the option to enroll in LTE study 77242113PSO2002 (NCT05364554). Participants who were not enrolled in LTE study were followed up for safety up to 4 weeks after the last dose of the study drug at Week 16.
- JNJ-77242113 100 mg BID: Participants with moderate to severe plaque psoriasis received JNJ-77242113 100 mg BID in morning and evening along with a matching placebo in morning to maintain the blind from Week 0 through Week 16. At Week 16 participants had the option to enroll in LTE study 77242113PSO2002 (NCT05364554). Participants who were not enrolled in LTE study were followed up for safety up to 4 weeks after the last dose of the study drug at Week 16.
Period: Overall Study
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Started | 43 | 43 | 43 | 41 | 43 | 42
Completed | 36 | 36 | 40 | 40 | 41 | 38
Not Completed | 7 | 7 | 3 | 1 | 2 | 4
Not completed — Lost to Follow-up | 1 | 3 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 2 | 3 | 1 | 1 | 2
Not completed — Other | 0 | 2 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID | Total
Number analyzed (Participants) | 43 | 43 | 43 | 41 | 43 | 42 | 255
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (14.7) | 44.5 (12.72) | 45.1 (11.08) | 45.7 (11.91) | 44.7 (14.11) | 42 (11.34) | 44.3 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 16 | 11 | 11 | 12 | 79
  Male | 25 | 32 | 27 | 30 | 32 | 30 | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 4 | 3 | 3 | 2 | 19
  Not Hispanic or Latino | 39 | 39 | 38 | 37 | 40 | 40 | 233
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 1 | 1 | 0 | 5
  Asian | 5 | 12 | 9 | 7 | 7 | 9 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Black or African American | 0 | 0 | 0 | 3 | 0 | 2 | 5
  White | 37 | 30 | 31 | 27 | 35 | 30 | 190
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 0 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 7 | 6 | 4 | 7 | 6 | 5 | 35
  France | 1 | 1 | 2 | 1 | 1 | 1 | 7
  Germany | 8 | 8 | 9 | 7 | 9 | 6 | 47
  Japan | 3 | 3 | 3 | 3 | 4 | 4 | 20
  Korea, South | 1 | 2 | 3 | 1 | 1 | 3 | 11
  Poland | 8 | 9 | 11 | 9 | 13 | 10 | 60
  Spain | 2 | 2 | 1 | 2 | 1 | 1 | 9
  Taiwan | 1 | 4 | 3 | 3 | 2 | 0 | 13
  United Kingdom | 2 | 0 | 0 | 0 | 0 | 1 | 3
  United States | 10 | 8 | 7 | 8 | 6 | 11 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved at Least 75 Percent (%) Improvement From Baseline in Psoriasis Area and Severity Index (PASI-75) at Week 16
Description: Percentage of participants who achieved PASI-75 score (greater than or equal to [>=] 75% improvement from baseline in PASI) at Week 16 was reported. The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed and scored separately for erythema, induration, and scaling, which were each rated on a scale of 0 to 4 (0=none, 1 = slight, 2 = moderate, 3 = severe and 4 = very severe) and extent of involvement from 0 (indicated no involvement) to 6 (90% - 100% involvement). The PASI produced a numeric total score that could range from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated greater severity of psoriasis. The baseline was defined as the closest measurement taken prior to or at the time of the first study drug administration date.
Time Frame: Baseline (Week 0), Week 16
Population: Full analysis set (FAS) included all randomized participants who received at least 1 administration of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 43 | 43 | 43 | 41 | 43 | 42
Percentage of participants | 9.3 | 37.2 | 58.1 | 51.2 | 65.1 | 78.6
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose versus (vs) placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

2. Secondary Outcome: Change From Baseline in PASI Total Score at Week 16
Description: Change from baseline in PASI total score at Week 16 was reported. The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed and scored separately for erythema, induration, and scaling, which were each rated on a scale of 0 to 4 (0=none, 1 = slight, 2 = moderate, 3 = severe and 4 = very severe) and extent of involvement from 0 (indicated no involvement) to 6 (90% - 100% involvement). The PASI produced a numeric total score that could range from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated greater severity of psoriasis. The baseline was defined as the closest measurement taken prior to or at the time of the first study drug administration date.
Time Frame: Baseline (Week 0), Week 16
Population: FAS included all randomized participants who received at least 1 administration of study intervention. Here, 'N' (overall number of participants analyzed) signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 40 | 37 | 41 | 40 | 42 | 39
Units on a scale | -3.59 (9.436) | -12.76 (8.050) | -14.56 (6.528) | -12.73 (8.021) | -13.99 (8.653) | -17.44 (8.356)
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

3. Secondary Outcome: Percentage of Participants Who Achieved at Least 90% Improvement From Baseline in PASI (PASI-90) at Week 16
Description: Percentage of participants who achieved PASI-90 score (>=90% improvement from baseline in PASI) at Week 16 was reported. The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed and scored separately for erythema, induration, and scaling, which were each rated on a scale of 0 to 4 (0 = none, 1 = slight, 2 = moderate, 3 = severe and 4 = very severe) and extent of involvement from 0 (indicated no involvement) to 6 (90% - 100% involvement). The PASI produced a numeric total score that could range from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated greater severity of psoriasis. The baseline was defined as the closest measurement taken prior to or at the time of the first study drug administration date.
Time Frame: Baseline (Week 0), Week 16
Population: FAS included all randomized participants who received at least 1 administration of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 43 | 43 | 43 | 41 | 43 | 42
Percentage of participants | 2.3 | 25.6 | 51.2 | 26.8 | 46.5 | 59.5
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

4. Secondary Outcome: Percentage of Participants Who Achieved 100% Improvement From Baseline in PASI (PASI-100) at Week 16
Description: Percentage of participants who achieved PASI-100 score (100% improvement from baseline in PASI) at Week 16 was reported. The PASI was a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body was divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed and scored separately for erythema, induration, and scaling, which were each rated on a scale of 0 to 4 (0=none, 1 = slight, 2 = moderate, 3 = severe and 4 = very severe) and extent of involvement from 0 (indicated no involvement) to 6 (90% - 100% involvement). The PASI produced a numeric total score that could range from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated greater severity of psoriasis. The baseline was defined as the closest measurement taken prior to or at the time of the first study drug administration date.
Time Frame: Baseline (Week 0), Week 16
Population: FAS included all randomized participants who received at least 1 administration of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 43 | 43 | 43 | 41 | 43 | 42
Percentage of participants | 0 | 11.6 | 25.6 | 9.8 | 23.3 | 40.5
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p = 0.021, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p = 0.038, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

5. Secondary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) at Week 16
Description: The IGA assesses participant's plaque psoriasis. Lesions were graded for induration, erythema and scaling, each using a 5 point scale. Induration: 0 = no evidence of plaque elevation, 1 = minimal plaque elevation, = 0.25 millimeters (mm); 2 = mild plaque elevation, = 0.5 mm; 3 = moderate plaque elevation, = 0.75 mm; 4 = severe plaque elevation, greater than (>) 1 mm; Erythema: 0 = no evidence of erythema, hyperpigmentation may be present, 1 = faint erythema, 2 = light red coloration, 3 = moderate red coloration, 4 = bright red coloration; Scaling: 0 = no evidence of scaling, 1 = minimal; occasional fine scale over less than 5% of the lesion, 2 = mild; fine scale dominates, 3 = moderate; coarse scale predominates, 4 = severe; thick, scale predominates. Final IGA score of psoriasis was based upon the average of induration, erythema and scaling scores assessed on a 5 point scale: cleared (0), minimal (1), mild (2), moderate (3), or severe (4). Higher score indicated more severe disease.
Time Frame: At Week 16
Population: FAS included all randomized participants who received at least 1 administration of study intervention.
Measure: Number; unit: Percentages of participants
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 43 | 43 | 43 | 41 | 43 | 42
Percentages of participants | 11.6 | 39.5 | 58.1 | 51.2 | 62.8 | 64.3
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

6. Secondary Outcome: Percentage of Participants Who Achieved an IGA Score of Cleared (0) at Week 16
Description: The IGA assesses participant's plaque psoriasis. Lesions were graded for induration, erythema and scaling, each using a 5 point scale. Induration: 0 = no evidence of plaque elevation, 1 = minimal plaque elevation, = 0.25 mm; 2 = mild plaque elevation, = 0.5 mm; 3 = moderate plaque elevation, = 0.75 mm; 4 = severe plaque elevation, >1 mm; Erythema: 0 = no evidence of erythema, hyperpigmentation may be present, 1 = faint erythema, 2 = light red coloration, 3 = moderate red coloration, 4 = bright red coloration; Scaling: 0 = no evidence of scaling, 1 = minimal; occasional fine scale over less than 5% of the lesion, 2 = mild; fine scale dominates, 3 = moderate; coarse scale predominates, 4 = severe; thick, scale predominates. Final IGA score of psoriasis was based upon the average of induration, erythema and scaling scores assessed on a 5 point scale: cleared (0), minimal (1), mild (2), moderate (3), or severe (4). A higher score indicated more severe disease.
Time Frame: At Week 16
Population: FAS included all randomized participants who received at least 1 administration of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 43 | 43 | 43 | 41 | 43 | 42
Percentage of participants | 0 | 16.3 | 34.9 | 14.6 | 27.9 | 45.2
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

7. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) at Week 16
Description: A BSA was commonly used measure of severity of skin disease. It was defined as the percentage of surface area of the body involved with the condition being assessed, (that is, plaque psoriasis). BSA was assessed using hand print method where the surface area of the participant's hand including the palm and all 5 digits was used as a guide to estimate 1% BSA. The baseline was defined as the closest measurement taken prior to or at the time of the first study drug administration date.
Time Frame: Baseline (Week 0) and Week 16
Population: FAS included all randomized participants who received at least 1 administration of study intervention. Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 40 | 37 | 41 | 40 | 42 | 39
Percentage of BSA | -2.4 (16.51) | -11.9 (10.00) | -15.3 (11.41) | -13.3 (11.08) | -14.6 (14.03) | -21.0 (13.74)
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

8. Secondary Outcome: Change From Baseline in Psoriasis Symptoms and Signs Diary (PSSD) Symptoms Scores at Week 16
Description: Change from baseline in PSSD symptoms scores at Week 16 was reported. PSSD was a patient-reported outcome (PRO) questionnaire designed to measure severity of psoriasis symptoms and signs for the assessment of treatment benefit. PSSD was a self-administered PRO instrument that included 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Items were averaged on the daily symptom score when at least 3 items (>=50 percentage of 5 items) on these scales are answered. The average value was converted into 0-100 scoring, such that symptom score = average value*10, where, 0= least severe and 100= most severe. Higher score indicated more severe disease. The baseline was defined as the closest measurement taken prior to or at the time of the first study drug administration date.
Time Frame: Baseline (Week 0) and Week 16
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 40 | 37 | 41 | 40 | 42 | 39
Units on a scale | -0.8 (29.59) | -35.8 (29.22) | -36.7 (29.95) | -34.0 (29.19) | -29.4 (28.28) | -44.0 (31.22)
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

9. Secondary Outcome: Change From Baseline in PSSD Signs Score at Week 16
Description: Change from baseline in PSSD sign scores at Week 16 was reported. PSSD was a PRO questionnaire designed to measure severity of psoriasis symptoms and signs for assessment of treatment benefit. PSSD was a self-administered PRO instrument that included 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Items were averaged on the daily sign score when at least 3 items (>=50 percentage of 6 items) on these scales are answered. The average value was converted into 0-100 scoring, such that sign score = average value*10, where, 0= least severe and 100= most severe. Higher score indicated more severe disease. The baseline was defined as the closest measurement taken prior to or at the time of the first study drug administration date.
Time Frame: Baseline (Week 0) and Week 16
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 40 | 37 | 41 | 40 | 42 | 39
Units on a scale | -6.2 (22.38) | -38.6 (27.55) | -42.7 (28.70) | -41.8 (27.78) | -41.9 (28.65) | -51.1 (26.01)
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

10. Secondary Outcome: Percentage of Participants Who Achieved PSSD Symptoms Score Equal to (=) 0 at Week 16 Among Participants With a Baseline Symptoms Score Greater Than or Equal to (>=) 1
Description: The PSSD was a PRO questionnaire designed to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. PSSD was a self-administered PRO instrument that included 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Items were averaged on the daily symptom score when at least 3 items (>=50 percentage of 5 items) on these scales are answered. The average value was converted into 0-100 scoring, such that symptom score = average value*10, where, 0= least severe and 100= most severe. Higher score indicated more severe disease. The baseline was defined as the closest measurement taken prior to or at the time of the first study drug administration date.
Time Frame: Baseline (Week 0), Week 16
Population: Analysis population included all randomized participants who received at least 1 administration of study intervention and had baseline PSSD symptom score >=1.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 43 | 43 | 42 | 41 | 43 | 42
Percentage of participants | 0 | 16.3 | 23.8 | 17.1 | 27.9 | 26.2
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

11. Secondary Outcome: Percentage of Participants Who Achieved PSSD Sign Score = 0 at Week 16 Among Participants With a Baseline Sign Score >=1
Description: The PSSD was a PRO questionnaire designed to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. PSSD was a self-administered PRO instrument that included 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Items were averaged on the daily sign score when at least 3 items (>=50 percentage of 6 items) on these scales are answered. The average value was converted into 0-100 scoring, such that sign score = average value*10, where, 0= least severe and 100= most severe. Higher score indicated more severe disease. The baseline was defined as the closest measurement taken prior to or at the time of the first study drug administration date.
Time Frame: Baseline (Week 0) , Week 16
Population: Analysis population included all randomized participants who received at least 1 administration of study intervention and had baseline PSSD sign score >=1.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 43 | 43 | 43 | 41 | 43 | 42
Percentage of participants | 0 | 2.3 | 14.0 | 9.8 | 16.3 | 14.3
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p = 0.317, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p = 0.012, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p = 0.038, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p = 0.011, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

12. Secondary Outcome: Percentage of Participants Who Achieved a Dermatological Life Quality Index (DLQI) of 0 or 1 at Week 16 Among Participants With Baseline DLQI Score Greater Than (>) 1
Description: The DLQI was a dermatology specific health-related quality of life (HRQoL) instrument designed to assess the impact of the disease on a participant's HRQoL. It was a 10-item questionnaire that assesses HRQoL over the past week and in addition to evaluating overall HRQoL, could be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. Each question was scored on a 4-point scale of 0 to 3 (0 = not at all, 1 = a little; 2 = a lot; or 3 = very much, where higher score indicated more impact on QoL). The total score was sum of scores from all 10 questions and it ranged from 0 (not at all) to 30 (very much), with a higher score indicating greater impact on HRQoL. The baseline was defined as the closest measurement taken prior to or at the time of the first study drug administration date.
Time Frame: Baseline (Week 0), Week 16
Population: Analysis population included all randomized participants who received at least 1 administration of study intervention and had baseline DLQI score >1.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 41 | 43 | 43 | 40 | 43 | 41
Percentage of participants | 2.4 | 27.9 | 37.2 | 30.0 | 55.8 | 43.9
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

13. Secondary Outcome: Change From Baseline in Domain Scores of the Patient-Reported Outcomes Measurement Information System (PROMIS-29) at Week 16
Description: PROMIS-29, 29-item generic HRQoL survey, assesses each 7 PROMIS domains (depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; ability to participate in social roles and activities) with 4 questions and pain intensity. Questions ranked on 5-point Likert Scale (1=never, 2=rarely, 3=sometimes, 4=often and 5=always). Pain intensity was rated on 11-point scale (0=no pain; 10=worst imaginable pain). Higher score= worst pain. Each domain included 4 items, plus a single pain intensity item totaling 29 items. Raw score of each PROMIS domain was converted into a standardized score with mean of 50; standard deviation (SD) of 10 (T-Score). Higher PROMIS T-score=more of concept being measured i.e. higher scores in anxiety, depression, fatigue, pain interference, sleep disturbance= worse symptoms, higher scores in physical function, social roles= better functioning. Baseline: closest measurement taken prior to/at the time of first study drug administration date.
Time Frame: Baseline (Week 0) and Week 16
Population: FAS included all randomized participants who received at least 1 administration of study intervention. Here 'N' (overall number of participants analyzed) referred to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 40 | 37 | 41 | 40 | 42 | 39
Units on a scale
  Physical Function | -1.04 (5.929) | 2.30 (6.060) | 5.81 (6.896) | 4.55 (7.789) | 3.10 (7.325) | 5.81 (8.408)
  Anxiety | -2.36 (7.971) | -3.98 (8.789) | -5.27 (8.026) | -5.27 (6.787) | -4.70 (8.570) | -8.31 (9.693)
  Depression | -1.01 (6.238) | -3.09 (8.709) | -3.23 (6.576) | -1.96 (6.569) | -2.62 (7.465) | -3.67 (8.912)
  Fatigue | -0.76 (5.469) | -2.44 (10.983) | -1.50 (7.801) | -3.09 (8.676) | -2.98 (7.818) | -3.75 (8.409)
  Sleep Disturbance | 0.14 (6.099) | -1.89 (5.859) | -3.45 (7.947) | -4.36 (6.041) | -1.04 (5.995) | -3.19 (5.705)
  Social Roles and Activities | 0.99 (8.393) | 4.31 (9.035) | 4.82 (8.511) | 5.39 (10.908) | 5.78 (7.538) | 7.73 (9.607)
  Pain Interference | 0.09 (7.819) | -6.79 (9.038) | -7.41 (9.867) | -7.18 (7.956) | -3.98 (7.889) | -9.56 (8.668)
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Physical Function; Test type: Superiority; p = 0.002, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Physical Function; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Physical Function; Test type: Superiority; p = 0.002, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Physical Function; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Physical Function; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 6: Comparison: Placebo vs JNJ-77242113 25 mg QD; Anxiety; Test type: Superiority; p = 0.251, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 7: Comparison: Placebo vs JNJ-77242113 50 mg QD; Anxiety; Test type: Superiority; p = 0.087, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 8: Comparison: Placebo vs JNJ-77242113 25 mg BID; Anxiety; Test type: Superiority; p = 0.205, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 9: Comparison: Placebo vs JNJ-77242113 100 mg QD; Anxiety; Test type: Superiority; p = 0.082, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 10: Comparison: Placebo vs JNJ-77242113 100 mg BID; Anxiety; Test type: Superiority; p = 0.010, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 11: Comparison: Placebo vs JNJ-77242113 25 mg QD; Depression; Test type: Superiority; p = 0.357, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 12: Comparison: Placebo vs JNJ-77242113 50 mg QD; Depression; Test type: Superiority; p = 0.222, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 13: Comparison: Placebo vs JNJ-77242113 25 mg BID; Depression; Test type: Superiority; p = 0.987, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 14: Comparison: Placebo vs JNJ-77242113 100 mg QD; Depression; Test type: Superiority; p = 0.390, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 15: Comparison: Placebo vs JNJ-77242113 100 mg BID; Depression; Test type: Superiority; p = 0.380, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 16: Comparison: Placebo vs JNJ-77242113 25 mg QD; Fatigue; Test type: Superiority; p = 0.349, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 17: Comparison: Placebo vs JNJ-77242113 50 mg QD; Fatigue; Test type: Superiority; p = 0.553, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 18: Comparison: Placebo vs JNJ-77242113 25 mg BID; Fatigue; Test type: Superiority; p = 0.318, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 19: Comparison: Placebo vs JNJ-77242113 100 mg QD; Fatigue; Test type: Superiority; p = 0.207, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 20: Comparison: Placebo vs JNJ-77242113 100 mg BID; Fatigue; Test type: Superiority; p = 0.117, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 21: Comparison: Placebo vs JNJ-77242113 25 mg QD; Sleep Disturbance; Test type: Superiority; p = 0.156, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 22: Comparison: Placebo vs JNJ-77242113 50 mg QD; Sleep Disturbance; Test type: Superiority; p = 0.019, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 23: Comparison: Placebo vs JNJ-77242113 25 mg BID; Sleep Disturbance; Test type: Superiority; p = 0.004, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 24: Comparison: Placebo vs JNJ-77242113 100 mg QD; Sleep Disturbance; Test type: Superiority; p = 0.228, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 25: Comparison: Placebo vs JNJ-77242113 100 mg BID; Sleep Disturbance; Test type: Superiority; p = 0.034, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 26: Comparison: Placebo vs JNJ-77242113 25 mg QD; Social Roles and Activities; Test type: Superiority; p = 0.197, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 27: Comparison: Placebo vs JNJ-77242113 50 mg QD; Social Roles and Activities; Test type: Superiority; p = 0.107, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 28: Comparison: Placebo vs JNJ-77242113 25 mg BID; Social Roles and Activities; Test type: Superiority; p = 0.606, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 29: Comparison: Placebo vs JNJ-77242113 100 mg QD; Social Roles and Activities; Test type: Superiority; p = 0.004, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 30: Comparison: Placebo vs JNJ-77242113 100 mg BID; Social Roles and Activities; Test type: Superiority; p = 0.005, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 31: Comparison: Placebo vs JNJ-77242113 25 mg QD; Pain Interference; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 32: Comparison: Placebo vs JNJ-77242113 50 mg QD; Pain Interference; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 33: Comparison: Placebo vs JNJ-77242113 25 mg BID; Pain Interference; Test type: Superiority; p = 0.005, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 34: Comparison: Placebo vs JNJ-77242113 100 mg QD; Pain Interference; Test type: Superiority; p = 0.010, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 35: Comparison: Placebo vs JNJ-77242113 100 mg BID; Pain Interference; Test type: Superiority; p < 0.001, Mixed-Effect Model Repeated Measure — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

14. Secondary Outcome: Percentage of Participants Who Achieved at Least a 5-point Improvement From Baseline in Each PROMIS-29 Domain at Week 16
Description: PROMIS-29, 29-item generic HRQoL survey, assesses each 7 PROMIS domains (depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; ability to participate in social roles and activities) with 4 questions and pain intensity. Questions ranked on 5-point Likert Scale (1=never, 2=rarely, 3=sometimes, 4=often, 5=always). Pain intensity was rated on 11-point scale (0=no pain; 10=worst imaginable pain). Higher score=worst pain. Each domain includes 4 items, plus a single pain intensity item totaling 29 items. Raw score of each PROMIS domain was converted into a standardized score with mean of 50; SD of 10 (T-Score). Higher PROMIS T-score= more of the concept being measured i.e. higher scores in anxiety, depression, fatigue, pain interference and sleep disturbance) indicated worse symptoms, higher scores in physical function and social roles= better functioning. Baseline: closest measurement taken prior to/at the time of first study drug administration date.
Time Frame: Baseline (Week 0), Week 16
Population: FAS included all randomized participants who received at least 1 administration of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 43 | 43 | 43 | 41 | 43 | 42
Percentage of participants
  Physical Function | 11.6 | 23.3 | 41.9 | 36.6 | 37.2 | 40.5
  Anxiety | 30.2 | 32.6 | 44.2 | 53.7 | 41.9 | 54.8
  Depression | 23.3 | 27.9 | 34.9 | 26.8 | 32.6 | 35.7
  Fatigue | 18.6 | 20.9 | 23.3 | 41.5 | 25.6 | 42.9
  Sleep Disturbance | 16.3 | 23.3 | 32.6 | 43.9 | 23.3 | 38.1
  Social Roles and Activities | 23.3 | 30.2 | 46.5 | 56.1 | 44.2 | 57.1
  Pain Interference | 20.9 | 46.5 | 55.8 | 51.2 | 41.9 | 64.3
Statistical Analysis 1: Comparison: Placebo vs JNJ-77242113 25 mg QD; Physical Function; Test type: Superiority; p = 0.160, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 2: Comparison: Placebo vs JNJ-77242113 50 mg QD; Physical Function; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 3: Comparison: Placebo vs JNJ-77242113 25 mg BID; Physical Function; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 4: Comparison: Placebo vs JNJ-77242113 100 mg QD; Physical Function; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 5: Comparison: Placebo vs JNJ-77242113 100 mg BID; Physical Function; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 6: Comparison: Placebo vs JNJ-77242113 25 mg QD; Anxiety; Test type: Superiority; p = 0.818, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 7: Comparison: Placebo vs JNJ-77242113 50 mg QD; Anxiety; Test type: Superiority; p = 0.179, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 8: Comparison: Placebo vs JNJ-77242113 25 mg BID; Anxiety; Test type: Superiority; p = 0.030, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 9: Comparison: Placebo vs JNJ-77242113 100 mg QD; Anxiety; Test type: Superiority; p = 0.267, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 10: Comparison: Placebo vs JNJ-77242113 100 mg BID; Anxiety; Test type: Superiority; p = 0.022, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 11: Comparison: Placebo vs JNJ-77242113 25 mg QD; Depression; Test type: Superiority; p = 0.620, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 12: Comparison: Placebo vs JNJ-77242113 50 mg QD; Depression; Test type: Superiority; p = 0.240, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 13: Comparison: Placebo vs JNJ-77242113 25 mg BID; Depression; Test type: Superiority; p = 0.710, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 14: Comparison: Placebo vs JNJ-77242113 100 mg QD; Depression; Test type: Superiority; p = 0.341, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 15: Comparison: Placebo vs JNJ-77242113 100 mg BID; Depression; Test type: Superiority; p = 0.204, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 16: Comparison: Placebo vs JNJ-77242113 25 mg QD; Fatigue; Test type: Superiority; p = 0.786, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 17: Comparison: Placebo vs JNJ-77242113 50 mg QD; Fatigue; Test type: Superiority; p = 0.597, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 18: Comparison: Placebo vs JNJ-77242113 25 mg BID; Fatigue; Test type: Superiority; p = 0.023, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 19: Comparison: Placebo vs JNJ-77242113 100 mg QD; Fatigue; Test type: Superiority; p = 0.438, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 20: Comparison: Placebo vs JNJ-77242113 100 mg BID; Fatigue; Test type: Superiority; p = 0.017, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 21: Comparison: Placebo vs JNJ-77242113 25 mg QD; Sleep Disturbance; Test type: Superiority; p = 0.419, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 22: Comparison: Placebo vs JNJ-77242113 50 mg QD; Sleep Disturbance; Test type: Superiority; p = 0.080, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 23: Comparison: Placebo vs JNJ-77242113 25 mg BID; Sleep Disturbance; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 24: Comparison: Placebo vs JNJ-77242113 100 mg QD; Sleep Disturbance; Test type: Superiority; p = 0.421, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 25: Comparison: Placebo vs JNJ-77242113 100 mg BID; Sleep Disturbance; Test type: Superiority; p = 0.025, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 26: Comparison: Placebo vs JNJ-77242113 25 mg QD; Social Roles and Activities; Test type: Superiority; p = 0.470, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 27: Comparison: Placebo vs JNJ-77242113 50 mg QD; Social Roles and Activities; Test type: Superiority; p = 0.023, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 28: Comparison: Placebo vs JNJ-77242113 25 mg BID; Social Roles and Activities; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 29: Comparison: Placebo vs JNJ-77242113 100 mg QD; Social Roles and Activities; Test type: Superiority; p = 0.040, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 30: Comparison: Placebo vs JNJ-77242113 100 mg BID; Social Roles and Activities; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 31: Comparison: Placebo vs JNJ-77242113 25 mg QD; Pain Interference; Test type: Superiority; p = 0.013, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 32: Comparison: Placebo vs JNJ-77242113 50 mg QD; Pain Interference; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 33: Comparison: Placebo vs JNJ-77242113 25 mg BID; Pain Interference; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 34: Comparison: Placebo vs JNJ-77242113 100 mg QD; Pain Interference; Test type: Superiority; p = 0.038, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not
Statistical Analysis 35: Comparison: Placebo vs JNJ-77242113 100 mg BID; Pain Interference; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Dose response assessment was adjusted for multiplicity. Pairwise comparisons between each dose vs placebo were not

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Event (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation where participants administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or resulted in congenital anomaly/birth defect. TEAE was defined as any event that occurred at or after the initial administration of study agent.
Time Frame: From Week 0 through Week 20
Population: The safety analyses set included all randomized participants who received at least 1 administration of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
Number analyzed (Participants) | 43 | 43 | 43 | 41 | 43 | 42
Participants
  TEAEs | 22 | 20 | 26 | 20 | 19 | 26
  TESAEs | 0 | 0 | 1 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: From Week 0 through Week 20
Description: The safety analyses set included all randomized participants who received at least 1 administration of study intervention.
Arm/Group | Placebo | JNJ-77242113 25 mg QD | JNJ-77242113 50 mg QD | JNJ-77242113 25 mg BID | JNJ-77242113 100 mg QD | JNJ-77242113 100 mg BID
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/43 | 0/41 | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 1/43 | 0/41 | 2/43 | 0/42
Other Adverse Events (participants affected / at risk) | 10/43 | 10/43 | 15/43 | 12/41 | 8/43 | 10/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | JNJ-77242113 25 mg QD (N=43) | JNJ-77242113 50 mg QD (N=43) | JNJ-77242113 25 mg BID (N=41) | JNJ-77242113 100 mg QD (N=43) | JNJ-77242113 100 mg BID (N=42)
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infected Cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | JNJ-77242113 25 mg QD (N=43) | JNJ-77242113 50 mg QD (N=43) | JNJ-77242113 25 mg BID (N=41) | JNJ-77242113 100 mg QD (N=43) | JNJ-77242113 100 mg BID (N=42)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 4 | 2 | 1 | 1
Covid-19 (Infections and infestations) | 5 | 5 | 3 | 8 | 2 | 4
Nasopharyngitis (Infections and infestations) | 2 | 1 | 8 | 3 | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT05223868/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT05223868/SAP_001.pdf